CLINICAL TRIAL: NCT02096250
Title: Iron Absorption From Wheat Flour in Haiti
Brief Title: Iron Absorption in Haiti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Principal Investigator, Isabelle Aeberli, PhD, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: EK 2013-N43
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — Fe(III)-EDTA; ferrous fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NaFeEDTA (Experimental): NaFeEDTA
  Interventions: Other: NaFeEDTA
- Ferrous fumarate (Experimental): Ferrous fumarate
  Interventions: Other: Ferrous fumarate
- NaFeEDTA + ferrous fumarate (Experimental): NaFeEDTA + ferrous fumarate
  Interventions: Other: NaFeEDTA + ferrous fumarate

INTERVENTIONS:
Other: NaFeEDTA
  Arms: NaFeEDTA
Other: Ferrous fumarate
  Arms: Ferrous fumarate
Other: NaFeEDTA + ferrous fumarate
  Arms: NaFeEDTA + ferrous fumarate

SUMMARY:
The government of Haiti plans to introduce a flour fortification program. The aim of the project it to inform the authorities on the most suitable iron compound for this fortification program. For this purpose, iron absorption from wheat flour using different iron compounds will be investigated.

ELIGIBILITY:
Mother-child pairs will be recruited!

Inclusion criteria for mothers :

* Women of reproductive age (18 to 45 years)
* Generally healthy
* Consenting to study participation

Exclusion criteria for mothers :

* Pregnancy or lactation
* Weight >65 kg
* Chronic illnesses which may influence iron absorption
* Severe anemia (Hb<10 g/dl)

Inclusion criteria for children:

* Age 4 years +/- 12 months
* Generally healthy

Exclusion criteria for children :

* Severe anemia (Hb<10 g/dl)
* Weight for height < -2 Z scores (wasting)
* Height of age < -2 Z score (stunting)

Furthermore, the following exclusion criteria apply to both mothers and children :

* Chronic illnesses or medication which may influence iron absorption (will be judged by investigator)
* Consumption of vitamin or mineral supplement (unless they agree to discontinue using them two weeks before beginning of the study until the las visit)
* Allergies or intolerances relevant to the test meal (gluten)
* Blood donation or major blood losses during the 2 months prior to the study
* Illness during the 4 weeks prior to the study (will be judged by investigator)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Iron absorption | 14 days after test meal consumption

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Aeberli, PhD, Principal Investigator — ETH Zurich (Switzerland)
Locations (1):
- Ministère de la Santé Publique et de la Population, Port-au-Prince, Haiti